CLINICAL TRIAL: NCT03616431
Title: Prospective Observational Study of Prevalence, Assessment and Treatment of Pancreatic Insufficiency in Patients With Pancreatic Malignancies
Brief Title: Pancreatic Cancer Dietary Assessment Study
Acronym: PanDA
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Pancreatic Cancer UK (Other)
Responsible Party: Sponsor
Other Study IDs: 15_DOG03_309
Record Dates: First submitted 2018-05-08; First posted 2018-08-06 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Neoplasm; Pancreas Adenocarcinoma; Well-Differentiated Neuroendocrine Carcinoma; Malignant Neoplasm of Pancreas
Keywords: Pancreatic malignancy; Pancreatic enzyme insufficiency; Pancreatic enzyme replacement therapy; Pancreatic-kit breath test
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Demographic cohort: A prospective cross-sectional assessment of the prevalence of PEI-related symptoms in up to n=150 patients with pancreatic malignancy.
- Diagnosis cohort: A sub-set (up to n=50) of the Demographic cohort patients will be tested to elucidate the most efficient diagnostic panel for PEI in pancreatic malignancy.
  An extra assessment for PEI diagnosis consisting of a breath test (Pancreo-KIT breath test) will be carried out during the following 1-2 weeks after the first appointment (which takes around six hours to complete and involves the administration of bread spread with 13C butter followed by collection of the patient's breath in small plastic vials at timed intervals. The vials will subsequently be analyzed for 13C quantity; details in Appendix 6). Following these diagnostic tests, patients will complete an "acceptability questionnaire" to assess their opinion regarding the burden that these diagnostic tests may add.
  Interventions: Diagnostic Test: Pancreo-KIT breath test
- Follow-up cohort: Validation of the diagnostic panel designed and tested in Step-1 of this study and evaluation of dietician intervention (including Pancreatic Enzyme Replacement Therapy; PERT) and its impact in weight loss, symptom evolution, chemotherapy receiving rate, quality of life and overall survival.

INTERVENTIONS:
Diagnostic Test: Pancreo-KIT breath test — Pancreo-Kit (Isomed Pharma, Madrid, Spain) is a breath test devised to measure Pancreatic Enzyme Insufficiency. It is a non-invasive method to obtain information about the digestion of consumed lipids; this in turn is informative about the exocrine enzyme activity of the pancreas (specifically pancreatic lipase). This kit is manufactured to EC directive 98/79/EEC and carries the CE mark.
  The test is based on measurement of 13C which is a stable naturally occurring environmental isotope of carbon with a nucleus containing 6 protons and 7 neutrons (note, it is not radioactive).
  Groups: Diagnosis cohort

SUMMARY:
This is a prospective observational study which aims to evaluate;

The prevalence of pancreatic insufficiency in patients with pancreatic malignancies (adenocarcinoma and neuroendocrine tumours).

The most appropriate diagnostic strategy. The impact that an adequate diagnosis and treatment may have on patients' outcome.

DETAILED DESCRIPTION:
Patients will prospectively receive a full nutritional assessment, pancreatic enzyme insufficiency (PEI) diagnosis and dietician education. This assessment will be performed as an outpatient in parallel with the medical oncology team, by the research dietician. This study will be performed in two steps (summarized in Figure 2);

Step-1 | A prospective cross-sectional assessment of the prevalence of PEI-related symptoms in up to n=150 patients with pancreatic malignancy (this will be termed 'the demographic cohort'). A sub-set of these patients (n=50) will be tested to elucidate the most efficient diagnostic panel for PEI in pancreatic malignancy (this will be termed 'the diagnosis cohort').

Step-2 | A prospective longitudinal validation of the diagnostic panel designed and tested in Step-1 and evaluation of dietician intervention (including PERT) and its impact in weight loss, symptom evolution, chemotherapy receiving rate, Quality of Life and overall survival (this will be termed 'the follow-up cohort' and will include up to n=50 patients).

All patients included in both steps will have a full nutritional assessment at baseline, and PERT treatment (as per standard of care if considered appropriate). Patients in the follow-up cohort will be reviewed (at least every 3 months for a maximum of 6 months since study entry) by dietician for further intervention and assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically/cytologically-proven or clinically-suspected (by specialist MDT) pancreatic malignancy including pancreatic ductal adenocarcinoma or pancreatic NET.
* Patients to be seen in the Medical Oncology HPB and NET team clinic for assessment
* Age ≥18 years with no upper age limit
* Patients must be able to give informed consent; Written consent will be required for patients to be included within the diagnostic cohort Verbal consent only will be required for patients to be included within the demographic cohort and the follow-up cohort

Additional cohort-specific criteria;

* Patients will be recruited into three different cohorts with differing levels of participation (termed demographic, diagnostic and follow-up). Patients will not be recruited into the follow-up cohort until recruitment of both demographic and diagnosis cohorts are complete and the interim analysis has been performed.
* Demographic cohort | All patients referred for consideration of cancer treatment options will be eligible. Patients will need to give verbal informed consent.
* Diagnosis cohort | Patients who are already consented for being included into the demographic cohort and who will be attending at least to one follow-up appointment and are considered to be fit enough for diagnostic assessment will be eligible. Patients will need to give written informed consent.
* Follow-up cohort | All patients referred for consideration of options of cancer treatment will be included; patients with a minimum of 3 months of follow-up will be included in the final analysis. Patients will need to give verbal informed consent.

Exclusion Criteria:

- As long as the inclusion criteria are fulfilled, there are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically/cytologically-proven or clinically-suspected (by specialist MDT) pancreatic malignancy including pancreatic ductal adenocarcinoma or pancreatic NET.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Determine prevalence of pancreatic enzyme insufficiency in patients with pancreatic neoplasms. | 2 years
  Prevalence will be given as a percentage of all patients with pancreatic neoplasms with evidence of pancreatic enzyme insufficiency

SECONDARY OUTCOMES:
To determine the prevalence of PEI-related symptoms at first oncological referral. | 1 year
  Percentage of patients with documented biochemical evidence of pancreatic enzyme insufficiency with related symptoms
To evaluate nutritional status of patients at the time of oncological referral (using a panel of 'standard of care' blood tests parameters). | 1 year
  Using defined dietetic endpoints
To assess the feasibility of performing the PEI breath test and the fecal elastase-1 measurement. | 1 year
  Described as a percentage of successful tests completed by patients
To assess, using the "acceptability questionnaire" (developed specifically for this study), the acceptability of these investigations by patients. | 1 year
  To quantify acceptability on a pre-defined score for each of the tests.
To identify, through semi structured interviews and thematic analysis, diet-related themes of interest in a subset of patients involved in this study | 1 year
  Themes will be described in a semi-quantitative report arising from the interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Juan W Valle, Professor, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carnie LE, Lamarca A, Vaughan K, Kapacee ZA, McCallum L, Backen A, Barriuso J, McNamara MG, Hubner RA, Abraham M, Valle JW. Prospective observational study of prevalence, assessment and treatment of pancreatic exocrine insufficiency in patients with inoperable pancreatic malignancy (PANcreatic cancer Dietary Assessment (PanDA): a study protocol. BMJ Open. 2021 May 13;11(5):e042067. doi: 10.1136/bmjopen-2020-042067. PMID 33986039
- See also: HRA summary of results link — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/panda-pancreatic-cancer-dietary-assessment-study-2/